CLINICAL TRIAL: NCT00901186
Title: A Randomized, Open Label, Multicenter, Laser-controlled Phase II Study Assessing the Efficacy and Safety of Ranibizumab (Intravitreal Injections) vs. Laser Treatment in Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: Efficacy and Safety of Ranibizumab (Intravitreal Injections) Versus Laser Treatment in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: RED-ES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DES01; 2009-010825-37 (EudraCT Number)
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2014-07

CONDITIONS: Diabetic Macular Edema; Visual Impairment
Keywords: Diabetic Macular Edema; Ranibizumab; Laser Treatment; Visual impairment
MeSH Terms: conditions — Vision Disorders | interventions — Ranibizumab

ARMS (2):
- RFB002 (Experimental): RFB002 0.5 mg was administered to the study eye with a single monthly intravitreal injection on day 1, day 30 and day 60. After day 90, if stable vision was not achieved, a monthly injection of RFB002 0.5 mg was administered until stable vision was achieved.
  Interventions: Drug: RFB002
- Laser photocoagulation (Active Comparator): At least one treatment of laser photocoagulation was applied on day 1. The maximum number of laser photocoagulation treatments was 4.
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Drug: RFB002 — 0.5 mg
  Other Names: Ranibizumab
  Arms: RFB002
Procedure: Laser photocoagulation
  Arms: Laser photocoagulation

SUMMARY:
This study will assess the efficacy and safety of ranibizumab (intravitreal injections) versus laser treatment in patients with visual impairment due to diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus 1 or 2, HbA1c < 11.0%, With: Clinically significant Diabetic Macular Edema in at least one eye.
2. Previous treatment with macular photocoagulation only should be considered if the investigator believes that the study eye may possibly benefit from additional photocoagulation.
3. Best corrected visual acuity score between 78 and 25 letters (Early Treatment Diabetic Retinopathy Study- ETDRS Chart - 4 meters).
4. Central foveal thickness >250µm (Optical Coherence Tomography).
5. Diabetes medication stable in the 3 months prior.

Exclusion Criteria:

In the study eye:

1. Active intraocular inflammation.
2. Any active infection.
3. History of uveitis.
4. Structural damage within 500 microns of the center of the macula.
5. Neovascularization of the iris.
6. Uncontrolled glaucoma in either eye (Intraocular Pressure > 24 mmHg).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Chair — Novartis
Locations (15):
- Spain (15):
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Novartis Investigative Site, San Cristóbal de La Laguna, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RFB002 | Laser Photocoagulation
Started | 40 | 43
Safety Set | 39 (One participant did not receive one intravitreal RFB002 injection.) | 43
Intent to Treat | 35 (Four treated participants did not have at least a baseline and one post-treatment BCVA.) | 38 (Five treated participants did not have at least a baseline and one post-treatment BCVA.)
Completed | 31 | 32
Not Completed | 9 | 11
Not completed — Lack of Efficacy | 0 | 1
Not completed — Abnormal laboratory values | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 2 | 4
Not completed — Administration problems | 0 | 1
Not completed — Protocol deviations | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RFB002 | Laser Photocoagulation | Total
Number analyzed (Participants) | 39 | 43 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.31 (8.94) | 65.47 (9.40) | 63.49 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: Visual acuity (VA) was assessed on the study eye during every study visit using best correction determined from protocol refraction. VA measurements were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters.
Time Frame: Baseline, 12 months
Population: Intent-to-treat (ITT): The ITT consisted of all randomized participants who received at least one intravitreal ranibizumab injection of one laser photocoagulation treatment for whom there was at least one baseline and one post-treatment BCVA value. Participants who had both Baseline and Month 12 BCVA values only were included in this analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 32 | 33
letters | 9.41 (9.15) | 5.79 (9.40)

2. Secondary Outcome: Percentage of Participants With Improvement in BCVA
Description: as for outcome 1
Time Frame: 12 months
Population: Intent-to-treat (ITT): The ITT consisted of all randomized participants who received at least one intravitreal ranibizumab injection of one laser photocoagulation treatment for whom there was at least one baseline and one post-treatment BCVA value.
Measure: Number; unit: Percentage of participants
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 35 | 38
Percentage of participants | 74.29 | 68.42

3. Secondary Outcome: Evolution of Mean Change From Baseline in BCVA by Study Visit
Description: as for outcome 1
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: ITT: The ITT consisted of all randomized participants who received at least one intravitreal ranibizumab injection of one laser photocoagulation treatment for whom there was at least one baseline and one post-treatment BCVA value. For each month, participants who had both the baseline and the study month BCVA values were included in the analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 35 | 38
letters
  Month 1 (n=34,38) | 4.56 (7.38) | 1.32 (7.99)
  Month 2 (n=31,38) | 4.61 (6.55) | 1.89 (8.04)
  Month 3 (n=33,38) | 6.24 (6.41) | 3.11 (7.83)
  Month 4 (n=33,37) | 6.33 (7.40) | 2.76 (8.66)
  Month 5 (n=31,37) | 7.03 (8.00) | 3.38 (8.95)
  Month 6 (n=33,35) | 7.61 (6.88) | 4.11 (7.65)
  Month 7 (n=33,33) | 7.91 (7.16) | 3.85 (7.97)
  Month 8 (n=32,34) | 8.00 (7.77) | 3.21 (7.75)
  Month 9 (n=32,33) | 8.44 (8.78) | 6.00 (9.81)
  Month 10 (n=31,32) | 7.32 (8.17) | 5.84 (9.14)
  Month 11 (n=32,32) | 7.69 (8.88) | 6.44 (8.32)
  Month 12 (n=32,33) | 9.41 (9.15) | 5.79 (9.40)

4. Secondary Outcome: Percentage of Participants With VA > 73 Letters With Ranibizumab (0.5 mg) vs Laser.
Description: VA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 35 | 38
Percentage of participants | 54.29 | 23.68

5. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) by Study Visit
Description: CRT was assessed by Optical Coherence Tomography (OCT).
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: ITT: The ITT consisted of all randomized participants who received at least one intravitreal ranibizumab injection of one laser photocoagulation treatment for whom there was at least one baseline and one post-treatment BCVA value. For each month, participants who had both the baseline and the study month CRT values were included in the analysis.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 35 | 38
micrometers
  Month 1 (n=33,37) | -50.18 (62.23) | -21.86 (82.86)
  Month 2 (n=31,38) | -69.52 (65.10) | -14.21 (66.95)
  Month 3 (n=33,37) | -80.64 (87.06) | -43.16 (89.74)
  Month 4 (n=33,38) | -81.79 (92.14) | -37.66 (83.29)
  Month 5 (n=30,37) | -77.77 (73.47) | -28.92 (91.51)
  Month 6 (n=33,34) | -93.73 (79.42) | -40.47 (100.12)
  Month 7 (n=33,35) | -92.76 (79.55) | -60.94 (110.05)
  Month 8 (n=32,34) | -92.41 (82.27) | -64.82 (110.05)
  Month 9 (n=32,34) | -81.59 (81.38) | -74.59 (112.75)
  Month 10 (n=31,31) | -83.32 (81.56) | -84.39 (102.79)
  Month 11 (n=32,33) | -98.03 (76.75) | -94.85 (114.67)
  Month 12 (n=32,33) | -76.28 (76.56) | -86.00 (115.53)

6. Secondary Outcome: Percentage of CRT Change From Baseline by Study Visit
Description: CRT was assessed by Optical Coherence Tomography (OCT).
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | RFB002 | Laser Photocoagulation
Number analyzed (Participants) | 35 | 38
Percentage change
  Month 1 (n=33,37) | -12.06 (15.16) | -3.01 (17.52)
  Month 2 (n=31,38) | -15.61 (13.90) | -2.20 (15.24)
  Month 3 (n=33,37) | -18.25 (17.09) | -7.97 (17.80)
  Month 4 (n=33,38) | -18.00 (17.93) | -6.99 (17.18)
  Month 5 (n=30,37) | -18.21 (15.68) | -6.39 (19.27)
  Month 6 (n=33,34) | -20.69 (15.85) | -8.55 (21.06)
  Month 7 (n=33,35) | -21.11 (15.68) | -12.50 (23.05)
  Month 8 (n=32,34) | -21.20 (16.43) | -13.02 (20.95)
  Month 9 (n=32,34) | -19.17 (17.95) | -15.68 (21.87)
  Month 10 (n=31,31) | -19.55 (17.34) | -17.24 (19.63)
  Month 11 (n=32,33) | -22.65 (15.85) | -19.04 (22.31)
  Month 12 (n=32,33) | -18.23 (16.66) | -16.59 (25.06)

ADVERSE EVENTS:
Arm/Group | RFB002 | Laser Photocoagulation
Serious Adverse Events (participants affected / at risk) | 3/39 | 2/43
Other Adverse Events (participants affected / at risk) | 2/39 | 3/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RFB002 (N=39) | Laser Photocoagulation (N=43)
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RFB002 (N=39) | Laser Photocoagulation (N=43)
Pharyngitis (Infections and infestations) | 2 | 0
Cataract operation (Surgical and medical procedures) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.